CLINICAL TRIAL: NCT03494751
Title: Heart Monitoring Device After Acute Myocardium Infarction
Acronym: Monitor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5391/17
Record Dates: First submitted 2018-01-22; First posted 2018-04-11 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2018-04

CONDITIONS: Acute Myocardial Infarction
Keywords: Monitoring; Myocardial infarction; Clinical trial
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart Monitor (Experimental): We used the device (heart monitor) in the patients with myocardial infarction.
  Interventions: Device: Heart monitor
- No Heart Monitor (Active Comparator): No heart monitor device in the patients with myocardial infarction (control).
  Interventions: Device: No heart monitor

INTERVENTIONS:
Device: Heart monitor — Use of heart monitor device in the patients after acute myocardium infarct.
  Other Names: Heart monitor device
  Arms: Heart Monitor
Device: No heart monitor — Standard monitoring by nurses.
  Other Names: No heart monitor device
  Arms: No Heart Monitor

SUMMARY:
Verify the effectiveness of a Heart Monitor in preventing events in patients over 18 years after acute myocardial infarction in a clinical unit. Patients with neurological disease or congenital heart disease we excluded from the study.

DETAILED DESCRIPTION:
Heart Monitor can detect early intercurrences. Objective: To verify the effectiveness of a Heart Monitoring system in preventing events in patients after acute myocardial infarction. Methodology: This is a randomized clinical trial to be developed in a clinical unit and will include patients over 18 years , post-acute myocardial infarction who were transferred from the ICU emergency or hemodynamic to clinical unit. Patients with neurological disease or congenital heart disease will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years
* patients post-acute myocardial infarctium

Exclusion Criteria:

* patients with neurological disease
* patients with congenital heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Heart rhythm monitoring | One year
  Evaluating the effectiveness of a heart monitoring device in the prevention and detection of events in patients after acute myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: silvia goldmeier, Study Chair — Instituto de Cardiologia do Rio Grande do Sul